CLINICAL TRIAL: NCT00240968
Title: Evaluation of a Booster Dose of A/Vietnam/1203/04 (H5N1) Vaccine Administered at 6 Months to Healthy Adult Subjects After a Two Dose Schedule at 0 and 1 Months
Brief Title: H5 Booster After a Two Dose Schedule
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 05-0090
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2013-08-16 (Estimated); Status verified 2008-07

CONDITIONS: Influenza
Keywords: Avian influenza, vaccine, A/H5N1, sub-study
MeSH Terms: conditions — Influenza, Human; Influenza in Birds

ARMS (4):
- 3 (Experimental): Subjects will receive a single 45 mcg IM dose of the influenza A/H5N1 virus vaccine.
  Interventions: Biological: Inactivated Influenza A/H5N1 Vaccine (sanofi pasteur)
- 4 (Experimental): Subjects will receive a single 90 mcg IM dose of the influenza A/H5N1 virus vaccine.
  Interventions: Biological: Inactivated Influenza A/H5N1 Vaccine (sanofi pasteur)
- 1 (Experimental): Subjects will receive a single 7.5 mcg IM dose of the influenza A/H5N1 virus vaccine.
  Interventions: Biological: Inactivated Influenza A/H5N1 Vaccine (sanofi pasteur)
- 2 (Experimental): Subjects will receive a single 15 mcg IM dose of the influenza A/H5N1 virus vaccine.
  Interventions: Biological: Inactivated Influenza A/H5N1 Vaccine (sanofi pasteur)

INTERVENTIONS:
Biological: Inactivated Influenza A/H5N1 Vaccine (sanofi pasteur) — A monovalent subvirion H5N1 vaccine (HA of A/Vietnam/1203/04) provided in unit¿¿dose vials containing either 30-mcg/mL A/H5N1 HA or 90-mcg/mL A/H5N1 HA. Subjects will receive 1 of 4 dose levels of vaccine (7.5, 15, 45, or 90 mcg) administered intramuscularly.

SUMMARY:
The purpose of this study is to determine whether a third dose of vaccines containing A/Vietnam/1203/04 provides more immunity than two doses. Subjects who participate in this study will have participated in DMID protocol 04-063 involving the A/Vietnam/1203/04. In this study, each subject will be asked to receive a third dose of the H5 vaccine at the same level administered in protocol 04-063. Subjects will be asked to record oral temperature and any experienced side effects for 7 days following the vaccine. Study procedures will include up to 3 blood sample collections. Participants will be involved in study related procedures for up to 6 months.

DETAILED DESCRIPTION:
This study is linked to DMID protocols 04-063, 07-0022 and 08-0059. DMID Study 05-0090 is an extension study to DMID Study 04-063. Between March and May 2005, DMID Study 04-063 enrolled approximately 450 subjects at three study sites. Subjects were stratified by age and history of prior influenza vaccination for the 2004-2005 season, and randomly assigned to receive 2 doses of saline placebo (N=50) or 7.5, 15, 45, or 90 mcg of the influenza A/H5N1 virus vaccine (N=100/dose group) by IM injection. Approximately 6 months after receiving their second vaccination, subjects enrolled in DMID Study 04-063 will return to the clinic for their final study visit (Visit 6). After completing this visit, which includes collection of safety data and a 30-mL blood draw, the unblinded vaccine administrator will determine if the study subject received placebo or the influenza A/H5N1 vaccine. In the proposed extension study (DMID Study 05-0090), subjects who received the influenza A/H5N1 vaccine will be provided with information about DMID Study 05-0090 and asked if they are willing to receive a third dose of vaccine at the same dose level originally administered (i.e., those subjects originally receiving two doses of 7.5 mcg will receive a single booster dose of 7.5 mcg, those receiving two doses of 15 mcg will receive a single booster of 15 mcg, etc.). Subjects that provide informed consent and are eligible for DMID Study 05-0090 will be given a third dose of the vaccine at the same dose level they previously received by the unblinded vaccine administrator. Symptoms and signs will be assessed in the clinic for 15 to 30 minutes after inoculation, and the subjects will maintain a memory aid to record oral temperature and systemic and local adverse events (AEs) for 7 days after each immunization. Subjects will be encouraged to take their temperature around the same time each day. All subjects will receive a safety follow-up telephone call at 1 to 3 days to elicit any AE information and between 13 to 19 days after the vaccination to elicit any AE information and review the memory aid. Subjects will return to the clinic 28 (+/- 3) days after vaccination for assessment of AEs and concomitant medications, targeted physical examination (if indicated) and blood sample collection. During this follow-up visit, subjects who have been identified as "high responders" to the vaccine in the DMID 04-063 study will also be solicited to participate in a blood specimen collection substudy. Subjects will be provided with information about the substudy and asked if they would consent to have an additional 100 mL of blood drawn after the blood sample is collected for serum antibody assays. Refusal to consent for this substudy does not preclude subjects from continuing in the booster vaccine trial. At approximately Day 180 (6 months after booster vaccination), subjects will return to the clinic for a final immunogenicity blood sample collection and for follow-up, which may include a targeted physical examination (if indicated). The duration of the study treatment for each subject in this study will be about 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Previous recipient of inactivated Influenza A/H5N1 vaccine in study DMID 04-063.
* Male or nonpregnant female (as indicated by a negative urine pregnancy test immediately prior to vaccine administration) between the ages of 18 and 65 years, inclusive.
* Women of childbearing potential who are at risk of becoming pregnant must agree to practice adequate contraception (i.e., barrier method, abstinence, and licensed hormonal methods) for the entire study period.
* Is in good health, as determined by vital signs (heart rate, blood pressure, oral temperature), medical history and a targeted physical examination based on medical history.
* Able to understand and comply with planned study procedures.
* Provides informed consent prior to any study procedures and is available for all study visits.

In order to be eligible to participate in the blood specimen collection substudy, subjects must also meet the following additional inclusion criteria:

* Previously achieved a 4-fold or greater increase from baseline in GMT following the second immunization with A/H5N1 approximately 28 days after dose 2 of study DMID 04-063 (approximately Day 56).
* Agrees to the storage of clinical specimens for an indefinite period of time at a central laboratory for use in future research.

Exclusion Criteria:

* Received placebo in DMID Study 04-063.
* Known allergy to eggs or other components of the vaccine or latex.
* Has a positive urine pregnancy test prior to vaccination (if female of childbearing potential) or women who are breastfeeding.
* Is undergoing immunosuppression as a result of an underlying illness or treatment.
* Has or had a neoplastic disease diagnosed or treated within the last 5 years or any lifetime history of hematologic malignancy. Those participants with any history of benign basal cell carcinoma of the skin may participate.
* Is using oral or parenteral steroids, high-dose inhaled steroids (>800 micrograms/day of beclomethasone dipropionate or equivalent) or other immunosuppressive or cytotoxic drugs.
* Has a history of receiving immunoglobulin or other blood product within the 3 months prior to enrollment in this study.
* Has received any other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrollment in this study.
* Has an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses (this includes, but is not limited to: known chronic liver disease, significant renal disease, unstable or progressive neurological disorders, diabetes mellitus, and transplant recipients).
* Has a history of severe reactions following immunization with contemporary influenza virus vaccines.
* Has an acute illness, including an isolated oral temperature greater than 100.4 degrees F, within 1 week of vaccination.
* Received an experimental agent (vaccine, drug, biologic, device, blood product, or medication) within 1 month prior to enrollment in this study other than DMID 04-063, or expects to receive an experimental agent during the 7-month study period.
* Has a history of alcohol abuse or drug abuse (including chronic pain medication) in the last 5 years.
* Has any condition that would, in the opinion of the site investigator, place the subject at an unacceptable risk of injury or render the subject unable to meet the requirements of the protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2005-10; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects in each dose group achieving a serum neutralizing antibody titer of 1:40 against the influenza A/H5N1 virus. | Day 28 following booster immunization.
Adverse event (AE) or serious adverse event (SAE) information (solicited in-clinic and via memory aids, concomitant medications, and periodic targeted physical assessments). | Adverse Events will be collected through day 28. Serious Adverse Events will be collected throughout the study through day 180.

SECONDARY OUTCOMES:
Proportion of subjects in each group achieving a day 28 post boost titer that is a 4-fold or greater increase compared to the peak titer achieved after the first two doses of vaccine. | Day 28.
Geometric mean titer of serum neutralizing and HAI antibodies at 28 and 180 days following booster immunization. | Day 28 and 180.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - UCLA Center For Vaccine Research, Torrance, California
  - University of Maryland Baltimore, Baltimore, Maryland
  - University of Rochester Medical Center - Strong Memorial Hospital - Infectious Diseases, Rochester, New York

REFERENCES:
- [Result] Zangwill KM, Treanor JJ, Campbell JD, Noah DL, Ryea J. Evaluation of the safety and immunogenicity of a booster (third) dose of inactivated subvirion H5N1 influenza vaccine in humans. J Infect Dis. 2008 Feb 15;197(4):580-3. doi: 10.1086/526537. PMID 18237269